CLINICAL TRIAL: NCT04177160
Title: The Effects of Music on Autonomic Nervous System and Anxiety in Healthy Elderly and Persons With Subjective Cognitive Decline
Brief Title: The Effects of Music on ANS and Anxiety in Healthy Elderly and Persons With SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902035RINC
Record Dates: First submitted 2019-11-13; First posted 2019-11-26 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Dementia
Keywords: music; anxiety; autonomic nervous system; subjective cognition decline
MeSH Terms: conditions — Dementia; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCD subjects (Experimental): Patients were diagnosed with subjective cognition decline and referred by neurologists.
  Interventions: Behavioral: Music; Behavioral: White noise
- Healthy controls (Experimental): Voluntary healthy elderly recruited from the community.
  Interventions: Behavioral: Music; Behavioral: White noise

INTERVENTIONS:
Behavioral: Music — Subjects sit still and listen to preferred music for 5 minutes.
Behavioral: White noise — Subjects sit still and listen to white noise for 5 minutes.

SUMMARY:
Subjective cognition decline (SCD) is considered as a risk factor of dementia and associates not only with further cognition deterioration but with a higher anxiety level. Anxiety may lead to decreasing cognitive function and negative impacts on the well-being and quality of life. To avoid these consequences, reducing anxiety is an important step to treat SCD. To ease anxious emotions, music has been viewed as an effective, safe and easy alternative to medication. Thus, the purpose of this study is to investigate the effects of music on reducing the anxiety of the healthy elderly and SCD and further to compare the anxiety level between SCD and healthy controls.

DETAILED DESCRIPTION:
Single subject pretest-posttest design was used. 12 SCD subjects was recruited from the memory clinic and 12 healthy controls from the community. The anxiety level was assessed both by self-reports (State-Trait Anxiety Inventory and Visual Analogue Scale of Anxiety) and by objective measurements related to autonomic nervous system activities (heart rate variability and electrodermal activity). The participants underwent a memory task to induce anxiety. Next, preferred music and white noise were provided in random order. The anxiety level and the effects of music intervention between SCD and healthy controls will be further compared.

ELIGIBILITY:
Inclusion Criteria:

* able to read and write Mandarin
* the scores of the Montreal Cognitive Assessment (MoCA) ≥ 24

Exclusion Criteria:

* cognitive status was affected by psychic problems, neurological disease or other conditions
* people with auditory and visual impairments
* people with obesity (BMI ≥ 27) or diabetes mellitus.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 45 minutes
  Heart activity was transformed into low- and high-frequency power components, which represented sympathetic and parasympathetic system activities respectively. It is recorded by skin conductance sensors wearing on the 2nd to 4th finger. These sensors connect to ProComp2™ Biofeedback System to collect biofeedback data. The data is further calibrated and analyzed by CardioPro Infiniti software.
Skin conductance | 45 minutes
  Electrodermal activity related to sympathetic system response (sweating). It is recorded by skin conductance sensors wearing on the 2nd to 4th finger. These sensors connect to ProComp2™ Biofeedback System to collect biofeedback data. The data is further calibrated and analyzed by CardioPro Infiniti software.
Visual Analogue Scale of Anxiety | After each stimulus task and intervention: on the 10th, 15th, 20th, 25th, 35th and 40th minute.
  Participants reports their immediately subjective anxiety levels.

SECONDARY OUTCOMES:
Chinese version of state-trait anxiety inventory-trait version | Baseline
  A self-report regards to participants' usual emotional status and personal characteristic based on a 4-point Likert scale and consists of 20 questions. People who get higher scores are considered having more anxious personality.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jessen F, Amariglio RE, van Boxtel M, Breteler M, Ceccaldi M, Chetelat G, Dubois B, Dufouil C, Ellis KA, van der Flier WM, Glodzik L, van Harten AC, de Leon MJ, McHugh P, Mielke MM, Molinuevo JL, Mosconi L, Osorio RS, Perrotin A, Petersen RC, Rabin LA, Rami L, Reisberg B, Rentz DM, Sachdev PS, de la Sayette V, Saykin AJ, Scheltens P, Shulman MB, Slavin MJ, Sperling RA, Stewart R, Uspenskaya O, Vellas B, Visser PJ, Wagner M; Subjective Cognitive Decline Initiative (SCD-I) Working Group. A conceptual framework for research on subjective cognitive decline in preclinical Alzheimer's disease. Alzheimers Dement. 2014 Nov;10(6):844-52. doi: 10.1016/j.jalz.2014.01.001. Epub 2014 May 3. PMID 24798886